CLINICAL TRIAL: NCT02317718
Title: Serum Vitamin D Level in Subfertile Women and Its Association With Ovarian Reserve and IVF Outcome.
Brief Title: Serum Vitamin D Level and Its Association With Ovarian Reserve and IVF Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fakih IVF Fertility Center (Other)
Responsible Party: Principal Investigator, monika chawla, Specialist Reproductive Endocrinology and Infertility, Fakih IVF Fertility Center
Other Study IDs: VitD Study
Record Dates: First submitted 2014-12-09; First posted 2014-12-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: VITAMIN D Disorders
Keywords: serum vitamin D levels; IVF; ovarian reserve; 25 OHD3; pregnancy outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal vitamin D levels group: MORE THAN 20 NG/ML VITAMIN D LEVELS
  Interventions: Other: monitor reproductive outcome
- Deficient Vitamin D GROUP: LESS THAN 20 NG/ML LEVELS
  Interventions: Other: monitor reproductive outcome

INTERVENTIONS:
Other: monitor reproductive outcome

SUMMARY:
Vitamin D has a major play in bone and calcium metabolism. Vitamin D deficiency (below 20 ng/ml) has also been linked to adverse health outcomes such as malignancy, cardiovascular disease, immune functioning, and glucose metabolism. Recent data from retrospective and prospective trials have demonstrated contradictive results concerning the role of vitamin D in female reproduction and IVF outcome. Some studies have found that women deficient in vitamin D had lower ovarian reserve and significantly lower clinical pregnancy rates when compared to patients who were sufficient levels in vitamin D. Some studies also demonstrated that serum 25-OH-D3 levels correlates with antimullerian hormone (AMH) levels in women of advanced reproductive age. It may also have a role to play in endocrine dysfunction and abnormal folliculogenesis in polycystic ovaries .

The aim of this prospective cohort study including infertile women undergoing IVF treatment is to investigate the association between serum 25-OH- D3 levels and parametres of ovarian reserve (AMH, antral follicle count, number of oocytes collected) and clinical pregnancy and miscarriage rates .

DETAILED DESCRIPTION:
Vitamin D has a major play in bone and calcium metabolism. Vitamin D deficiency (below 20 ng/ml) has also been linked to adverse health outcomes such as malignancy, cardiovascular disease, immune functioning, and glucose metabolism. Recent data from retrospective and prospective trials have demonstrated contradictive results concerning the role of vitamin D in female reproduction and IVF outcome. Some studies have found that women deficient in vitamin D had lower ovarian reserve and significantly lower clinical pregnancy rates when compared to patients who were sufficient levels in vitamin D. Some studies also demonstrated that serum 25-OH-D3 levels correlates with antimullerian hormone (AMH) levels in women of advanced reproductive age. It may also have a role to play in endocrine dysfunction and abnormal folliculogenesis in polycystic ovaries .

The aim of this prospective cohort study including infertile women undergoing IVF treatment is to investigate the association between serum 25-OH- D3 levels and parametres of ovarian reserve (AMH, antral follicle count, number of oocytes collected) and clinical pregnancy and miscarriage rates .

ELIGIBILITY:
Inclusion Criteria:

* Subfertile women,
* Indication for IVF,
* 20-42 yrs of age.

Exclusion Criteria:

* Women on therapeutic supplementation for Vitamin D Deficiency,
* Recurrent high order implantation failure

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing IVF between 20-42 years of age
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 14 days post oocyte retrieval

SECONDARY OUTCOMES:
AMH (antimullerian hormone) Levels | day 2-3 of the index cycle
AFC (antral follicle count) | DAY 2-3 OF INDEX CYCLE
Number of oocytes retreived | Two weeks from the last menstrual period

CONTACTS AND LOCATIONS:
Locations (1):
- Fakihivf Fertiity Center, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

REFERENCES:
- [Background] Paffoni A, Ferrari S, Vigano P, Pagliardini L, Papaleo E, Candiani M, Tirelli A, Fedele L, Somigliana E. Vitamin D deficiency and infertility: insights from in vitro fertilization cycles. J Clin Endocrinol Metab. 2014 Nov;99(11):E2372-6. doi: 10.1210/jc.2014-1802. Epub 2014 Aug 14. PMID 25121462
- [Background] Polyzos NP, Anckaert E, Guzman L, Schiettecatte J, Van Landuyt L, Camus M, Smitz J, Tournaye H. Vitamin D deficiency and pregnancy rates in women undergoing single embryo, blastocyst stage, transfer (SET) for IVF/ICSI. Hum Reprod. 2014 Sep;29(9):2032-40. doi: 10.1093/humrep/deu156. Epub 2014 Jun 20. PMID 24951484
- [Result] Fabris A, Pacheco A, Cruz M, Puente JM, Fatemi H, Garcia-Velasco JA. Impact of circulating levels of total and bioavailable serum vitamin D on pregnancy rate in egg donation recipients. Fertil Steril. 2014 Dec;102(6):1608-12. doi: 10.1016/j.fertnstert.2014.08.030. Epub 2014 Sep 23. PMID 25256926
- See also: Impact of circulating levels of total and bioavailable serum vitamin D on pregnancy rate in egg donation recipients. Fabris A, Pacheco A, Cruz M, Puente JM, Fatemi H, Garcia-Velasco JA. Fertil Steril. 2014 Dec;102(6):1608-12. — http://www.ncbi.nlm.nih.gov/pubmed/25265402
- See also: Vitamin D Deficiency and Infertility: Insights From in vitro Fertilization Cycles. Paffoni A, Ferrari S, Viganò P, Pagliardini L, Papaleo E, Candiani M, Tirelli A, Fedele L, Somigliana E. J Clin Endocrinol Metab. 2014 N — http://www.ncbi.nlm.nih.gov/pubmed/25256926
- See also: Vitamin D deficiency and pregnancy rates in women undergoing single embryo, blastocyst stage, transfer (SET) for IVF/ICSI. Polyzos NP1, Anckaert E2, Guzman L3, — http://www.ncbi.nlm.nih.gov/pubmed/24951484